CLINICAL TRIAL: NCT02082210
Title: A Phase 1b/2 Study of Ramucirumab in Combination With LY2875358 in Patients With Advanced Cancer
Brief Title: A Study of Emibetuzumab in Combination With Ramucirumab (LY3009806) in Participants With Advanced Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15246; I4C-MC-JTBF (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Results first posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2018-03

CONDITIONS: Advanced Cancer; Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Hepatocellular Cancer; Renal Cell Carcinoma; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung | interventions — emibetuzumab; Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Emibetuzumab + Ramucirumab (Part A) (Experimental): Part A: Dose escalation (750mg, 2000mg) of Emibetuzumab administered intravenously (IV), on days 1 and 15 every 28 day cycle in combination with a fixed dose of 8mg/kg ramucirumab administered IV on Days 1 and 15 every 28 day cycle.
  Interventions: Drug: Emibetuzumab; Drug: Ramucirumab
- Emibetuzumab + Ramucirumab (Part B) (Experimental): Part B: Recommended 750mg Emibetuzumab dose from Part A to be administered IV, on days 1 and 15 every 28 day cycle in combination with a fixed dose of 8mg/kg ramucirumab administered IV on Days 1 and 15 every 28 day cycle.
  Interventions: Drug: Emibetuzumab; Drug: Ramucirumab

INTERVENTIONS:
Drug: Emibetuzumab — Administered Intravenously (IV)
  Other Names: LY2875358
Drug: Ramucirumab — Administered Intravenously (IV)
  Other Names: LY3009806; IMC-1121B

SUMMARY:
The purpose of this study is to find a recommended schedule and dose range for Emibetuzumab when given with ramucirumab that may be safely given to participants with cancer. In Part A of this study, escalating doses of Emibetuzumab will be given in combination with a fixed dose of ramucirumab to evaluate the safety of the combination. After a recommended schedule and dose range of Emibetuzumab and ramucirumab has been established, Part B of the study will confirm safety and to see how well certain tumors respond to the combination of study drugs. The average amount of time on study is expected to be about 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histological or cytological confirmed diagnosis of the following tumor types that is advanced and/or metastatic cancer and must be, in the judgment of the investigator, an appropriate participant for experimental therapy

  * Part A: Any type of solid tumor ("all comer")
  * Part B1: Gastric or Gastroesophageal Junction (GEJ) adenocarcinoma
  * Part B2: Hepatocellular cancer (excluding fibrolamellar carcinoma)
  * Part B3: Renal cell carcinoma (any histology)
  * Part B4: Non-small cell lung cancer (squamous or non-squamous)
* Have at least 1 measurable lesion outside of the central nervous system (CNS) whose presence is assessable using standard techniques by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* Availability of a tumor sample taken after progression on the most recent line of systemic tumor therapy or willing to undergo a tumor biopsy pre-study treatment.
* Have a performance status of ≤ 2 on the Eastern Cooperative Oncology Group (ECOG) scale in Part A and ≤ 1 on the ECOG scale in Part B.
* Have adequate organ function.
* Routine urinalysis showing ≤1+ protein or protein/creatinine ratio <0.5. For proteinuria ≥2+ or urine protein/creatinine ratio ≥0.5, 24-hour urine must be collected and the level must be <1 gram of protein in 24 hours for subject enrollment.
* Have discontinued all previous cancer therapies and any agents that have not received regulatory approval for any indication, for at least 21 days or 5 halflives prior to study enrollment, whichever is shorter, and recovered from the acute effects for therapy.
* Have an estimated life expectancy, in the judgment of the investigator, that will permit the participant to complete 8 weeks (2 cycles) of treatment.
* Males and females with reproductive potential: Must agree to use medically approved contraceptive precautions during the study and for at least 3 months following the last dose of study drug. Females with childbearing potential must have had a negative serum pregnancy test 7 days before the first dose of study drug and must not be breast-feeding.

Exclusion Criteria:

* Have serious pre-existing medical conditions (at the discretion of the investigator, such as severe acute or chronic medical condition or laboratory abnormality that may increase the risk associated with study participation).
* Have a history of hypertensive crisis or hypertensive encephalopathy or current poorly controlled hypertension despite standard medical management.
* Participant has experienced any arterial thromboembolic event (ATE), including myocardial infarction, unstable angina pectoris, cerebrovascular accident, or transient ischemic attack, within 6 months prior to receiving study drugs.
* Have a history of deep vein thrombosis, pulmonary embolism, or any other significant thromboembolic event during the 3 months prior to receiving study drugs.
* Are receiving therapeutic anticoagulation with warfarin, low-molecular weight heparin, or similar agents. Participants receiving prophylactic, low-dose anticoagulation therapy are eligible provided that they are on low-molecular weight heparin or oral factor Xa inhibitors.
* The participant is receiving chronic therapy with nonsteroidal anti-inflammatory drugs or other antiplatelet agents. Aspirin use at doses up to 325 mg/day is permitted.
* Have significant bleeding disorders, vasculitis, or had a significant bleeding episode from the gastrointestinal (GI) tract within 3 months prior to receiving study drugs.
* Have a history of GI perforation and/or fistulae within 6 months prior to receiving study drugs.
* Have congestive heart failure (CHF) New York Heart Association class ≥3 or symptomatic or poorly controlled cardiac arrhythmia.
* Have undergone major surgery within 28 days prior to receiving study drugs.
* Have a serious or nonhealing wound, peptic ulcer, or bone fracture within 28 days prior to receiving study drugs.
* Have a known active fungal, bacterial, and/or known viral infection. Hepatocellular cancer participants with chronic viral (B or C) hepatitis are eligible if they retain adequate liver function.
* Have liver cirrhosis with a Child-Pugh Stage of B or C.
* Have symptomatic CNS malignancy (with the exception of medulloblastoma) or metastasis.
* Have corrected QT (QTc) interval of >470 milliseconds on screening electrocardiogram (ECG).
* Have received previous treatment with ramucirumab or Emibetuzumab, except for participants enrolled in cohort B1 (Gastric or GEJ adenocarcinoma) and B4 (non- small cell lung cancer) who may have received previous ramucirumab treatment.
* Known hypersensitivity to any of the treatment components of ramucirumab or Emibetuzumab.
* Have a second primary malignancy that, in the judgment of the investigator and sponsor, may affect the interpretation of results.
* Are pregnant or breastfeeding.
* For Part B4 (non-small cell lung cancer) only:

  * The participant has radiologically documented evidence of major blood vessel invasion or encasement by cancer
  * Participants with a history of gross hemoptysis within 2 months prior to study treatment
  * The participant has radiographic evidence of intratumor cavitation, regardless of tumor histology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2014-03-07 (Actual); Primary Completion 2017-12-05 (Actual); Study Completion 2018-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Tennessee Oncology PLLC, Nashville, Tennessee

REFERENCES:
- See also: Click here for more information about this study: A Study of LY2875358 in Combination With Ramucirumab (LY3009806) in Participants With Advanced Cancer — https://www.lillytrialguide.com/en-US/studies/solid-tumor/JTBF#?postal=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part A: Completers are those who have completed one cycle of treatment. Part B: Completers are those who 1)Have measurable disease at baseline and at least one post-baseline tumor assessment; and 2) Were treated until PD or death, or discontinued due to an AE and completed the required follow-up.
Pre-assignment Details: Two part study, Part A with 2 cohorts (750 milligram (mg), 2000mg) & Part B with four tumor specific cohorts (gastric, hepatocellular carcinoma (HCC), renal cell carcinoma (RCC), non-small cell lung cancer (NSCLC)).
Groups:
- Part A - 750 mg Emibetuzumab: Participants received 8 milligram per kilogram (mg/kg) Ramucirumab followed by 750 mg Emibetuzumab given as intravenous (IV) infusion on days 1 and 15 of 28 days cycle.
- Part A - 2000 mg Emibetuzumab: Participants received 8 mg/kg Ramucirumab followed by 2000 mg Emibetuzumab given as intravenous (IV) infusion on days 1 and 15 of 28 days cycle.
- Part B - Gastric: Participants received 8 mg/kg Ramucirumab followed by 750mg Emibetuzumab given as intravenous (IV) infusion on days 1 and 15 of 28 days cycle.
- Part B - HCC; Part B - RCC; Part B - NSCLC: Participants received 8 mg/kg Ramucirumab followed by 750 mg Emibetuzumab given as intravenous (IV) infusion on days 1 and 15 of 28 days cycle.
Period: Overall Study
Arm/Group | Part A - 750 mg Emibetuzumab | Part A - 2000 mg Emibetuzumab | Part B - Gastric | Part B - HCC | Part B - RCC | Part B - NSCLC
Started | 3 | 3 | 16 | 45 | 15 | 15
Received at Least One Dose of Study Drug | 3 | 3 | 16 | 45 | 15 | 15
Completed | 3 | 3 | 13 | 39 | 12 | 13
Not Completed | 0 | 0 | 3 | 6 | 3 | 2
Not completed — Death | 0 | 0 | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 2 | 2
Not completed — Clinical Progression | 0 | 0 | 0 | 1 | 0 | 0
Not completed — No Post-Baseline Tumor Assesment | 0 | 0 | 1 | 2 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part A - 750 mg Emibetuzumab: Participants received 8 mg/kg Ramucirumab followed by 750 mg Emibetuzumab given as intravenous (IV) infusion on days 1 and 15 of 28 days cycle.
- Part B - HCC; Part B - RCC; Part B - NSCLC: Participants received 8 mg/kg Ramucirumab followed by 750mg Emibetuzumab given as intravenous (IV) infusion on days 1 and 15 of 28 days cycle.
- Total: Total of all reporting groups
Arm/Group | Part A - 750 mg Emibetuzumab | Part A - 2000 mg Emibetuzumab | Part B - Gastric | Part B - HCC | Part B - RCC | Part B - NSCLC | Total
Number analyzed (Participants) | 3 | 3 | 16 | 45 | 15 | 15 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (20.6) | 62.0 (13.5) | 62.6 (9.1) | 63.4 (9.5) | 63.1 (10.1) | 59.9 (8.6) | 62.0 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 4 | 11 | 3 | 6 | 27
  Male | 0 | 3 | 12 | 34 | 12 | 9 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: All participants with baseline ethnicity data.
  Participants
    number analyzed (Participants) | 3 | 3 | 16 | 39 | 15 | 14 | 90
    Hispanic or Latino | 0 | 0 | 1 | 3 | 2 | 0 | 6
    Not Hispanic or Latino | 3 | 3 | 15 | 36 | 13 | 14 | 84
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: All randomized participants with baseline race data.
  Participants
    number analyzed (Participants) | 3 | 3 | 15 | 43 | 14 | 14 | 92
    American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 1
    Asian | 0 | 0 | 0 | 7 | 0 | 2 | 9
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 1 | 1 | 3 | 0 | 1 | 6
    White | 3 | 2 | 14 | 32 | 14 | 11 | 76
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 16 | 45 | 15 | 15 | 97

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs)
Description: DLT is defined as an adverse event during Cycle1 that is possibly, probably, or definitely related to treatment with Emibetuzumab in combination with fixed regimen of Ramucirumab & fulfills any 1 of the following criterion using NCI CTCAE Version 4.03:
  Grade 3 non-hematological toxicity. Exceptions will be made for:Nausea, vomiting, diarrhea, constipation, or skin rash that persists for ≤3 days following appropriate supportive care intervention. Grade 3 hypertension in which systolic BP ≥160 mmHg and/or diastolic BP ≥100 mmHg persist <7 days after intensified antihypertensive therapy is initiated.
  Grade 4 hematological toxicity of ≥7 days duration.
  ≥Grade 3 thrombocytopenia with ≥Grade 2 bleeding.
  Any febrile neutropenia.
  Any other significant toxicity deemed by the primary investigator & Lilly clinical research personnel to be dose-limiting (eg, any toxicity that is possibly related to the study medication that requires the withdrawal of participant from study Cycle1).
Time Frame: Baseline through Cycle 1 (28 day cycle)
Population: All participants who received at least one dose of Emibetuzumab in Part A & Part B.
Measure: Count of Participants; unit: Participants
Groups:
- Part B - Gastric; Part B - HCC; Part B - RCC; Part B - NSCLC: Participants received 8 mg/kg Ramucirumab followed by 750 mg Emibetuzumab given as intravenous (IV) infusion on days 1 and 15 of 28 days cycle.
Arm/Group | Part A - 750 mg Emibetuzumab | Part A - 2000 mg Emibetuzumab | Part B - Gastric | Part B - HCC | Part B - RCC | Part B - NSCLC
Number analyzed (Participants) | 3 | 3 | 16 | 45 | 15 | 15
Participants | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Part B: Percentage of Participants Who Exhibit Complete Response (CR) or Partial Response (PR) [Overall Response Rate (ORR)]
Description: ORR is the percentage of participants achieving a best overall response (BOR) of complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR is defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR is defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. PD was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Baseline through Measured Progressive Disease or Death (Up to 17 months)
Population: All participants who received at least one dose of Emibetuzumab in Part B.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part B - Gastric | Part B - HCC | Part B - RCC | Part B - NSCLC
Number analyzed (Participants) | 16 | 45 | 15 | 15
percentage of participants | 6.3 [0 to 30] | 6.7 [0 to 20] | 0 [0 to 20] | 6.7 [0 to 30]

3. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Plasma Concentration (Cmax) of Emibetuzumab
Description: Pharmacokinetics (PK): Maximum Observed Plasma Concentration (Cmax) of Emibetuzumab.
Time Frame: Cycle 1: Day1 Predose, End of infusion, 3 Hours (h), 5h, 8h, 21h, 168h, 334h, 335h and 336h Post dose
Population: All participants who received at least one dose of Emibetuzumab and had evaluable PK samples in Part A & Part B.
  Per protocol analysis was performed per each dose irrespective of the study parts.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter (µg/mL)
Groups:
- All Parts - 750 mg Emibetuzumab: Participants received 8 mg/kg Ramucirumab followed by 750 mg Emibetuzumab given as intravenous (IV) infusion on days 1 and 15 of 28 days cycle.
- All Parts - 2000 mg Emibetuzumab: Participants received 8 mg/kg Ramucirumab followed by 2000 mg Emibetuzumab given as intravenous (IV) infusion on days 1 and 15 of 28 days cycle.
Arm/Group | All Parts - 750 mg Emibetuzumab | All Parts - 2000 mg Emibetuzumab
Number analyzed (Participants) | 24 | 3
Microgram per milliliter (µg/mL) | 210 (27) | 575 (33)

4. Secondary Outcome: Part B: Percentage of Participants Who Exhibit Stable Disease (SD) or Confirmed Response (CR) or Partial Response (PR) (Disease Control Rate [DCR])
Description: DCR is the proportion of participants who exhibit a SD or confirmed CR or PR relative to baseline. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the LD of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. SD was neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD for target lesions, no progression of non-target lesions, and no appearance of new lesions. Progressive disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Baseline through Measured Progressive Disease (Up to 17 months)
Population: All participants who received at least one dose of Emibetuzumab in Part B.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part B - Gastric | Part B - HCC | Part B - RCC | Part B - NSCLC
Number analyzed (Participants) | 16 | 45 | 15 | 15
percentage of participants | 50 [20 to 80] | 60 [40 to 70] | 46.7 [20 to 70] | 86.7 [60 to 100]

5. Secondary Outcome: Part B: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of first dose of study drug until first observation of objective (radiographically documented) PD as defined by RECIST v1.1 or death from any cause, whichever comes first. PD was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Baseline to Measured Progressive Disease or Death (Up to 17 Months)
Population: All participants who received at least one dose of Emibetuzumab in part B. Censored participants in Part B- Gastric = 4; Part B - HCC = 15; Part B - RCC = 7; Part - B NSCLC = 4;
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part B - Gastric | Part B - HCC | Part B - RCC | Part B - NSCLC
Number analyzed (Participants) | 16 | 45 | 15 | 15
months | 1.64 [1.35 to 4.60] | 5.42 [1.64 to 8.12] | 2.92 [1.18 to 7.39] | 6.57 [2.86 to 9.66]

6. Secondary Outcome: Pharmacokinetics: Area Under the Concentration-Time Curve (AUC) From Time Zero to Tlast of Emibetuzumab
Description: Pharmacokinetics: Area Under the Concentration-Time Curve (AUC) from time zero to tlast of Emibetuzumab.
Time Frame: Cycle 1: Day1 Predose, End of infusion, 3 Hours (h), 5h, 8h, 21h, 168h, 334h, 335h and 336h Post dose
Population: All participants who received at least one dose of Emibetuzumab and had evaluable PK samples in Part A & Part B.
  Per protocol, analysis was performed per each dose irrespective of study parts.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram * hour per milliliter(µg*h/mL)
Arm/Group | All Parts - 750 mg Emibetuzumab | All Parts - 2000 mg Emibetuzumab
Number analyzed (Participants) | 24 | 3
Microgram * hour per milliliter(µg*h/mL) | 29800 (26) | 86500 (25)

7. Secondary Outcome: Pharmacokinetics: Area Under the Concentration-Time Curve (AUC) of Ramucirumab
Description: Pharmacokinetics: Area Under the Concentration-Time Curve (AUC) of Ramucirumab.
Time Frame: Cycle 1: Day1 Predose, End of infusion, 3 Hours (h), 5h, 8h, 21h, 168h and 336h Post dose
Population: Noncompartmental PK parameters were not generated for Ramucirumab due to inadequate PK sampling.
Groups:
- All Parts - 750mg: Participants received 8 mg/kg Ramucirumab followed by 750 mg Emibetuzumab given as intravenous (IV) infusion on days 1 and 15 of 28 days cycle.
- All Parts - 2000mg: Participants received 8 mg/kg Ramucirumab followed by 2000 mg Emibetuzumab given as intravenous (IV) infusion on days 1 and 15 of 28 days cycle.
Arm/Group | All Parts - 750mg | All Parts - 2000mg
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants With Treatment Emergent Anti-Emibetuzumab Antibodies
Description: Participants were considered as treatment-emergent anti drug antibodies (TE ADA) positive if there is a ≥4-fold increase from baseline when ADAs were detected at baseline. If no ADAs were detected at baseline, TE ADA were defined as those with a titer 2 fold (1 dilution) greater than the minimum required dilution (MRD) of the screening assay (1:4 for anti-emibetuzumab antibodies).
Time Frame: Baseline through 46 Months
Population: All participants who received at least one dose of Emibetuzumab and had evaluable immunogenicity samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - 750 mg Emibetuzumab | Part A - 2000 mg Emibetuzumab | Part B - Gastric | Part B - HCC | Part B - RCC | Part B - NSCLC
Number analyzed (Participants) | 3 | 3 | 15 | 42 | 15 | 15
Participants | 0 | 0 | 0 | 3 | 0 | 0

9. Secondary Outcome: Pharmacokinetics: Maximum Observed Plasma Concentration (Cmax) of Ramucirumab
Description: Pharmacokinetics: Maximum Observed Plasma Concentration (Cmax) of Ramucirumab.
Time Frame: Cycle 1: Day1 Predose, End of infusion, 3 Hours (h), 5h, 8h, 21h, 168h and 336h Post dose
Population: Noncompartmental PK parameters were not generated for Ramucirumab due to inadequate PK sampling.
Arm/Group | All Parts - 750mg | All Parts - 2000mg
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Number of Participants With Treatment Emergent Anti-Ramucirumab Antibodies
Description: Participants were considered as treatment-emergent anti drug antibodies (TE ADA) positive if there is a ≥4-fold increase from baseline when ADAs were detected at baseline. If no ADAs were detected at baseline, TE ADA were defined as those with a titer 2 fold (1 dilution) greater than the minimum required dilution (MRD) of the screening assay (1:10 for anti-ramucirumab antibodies).
Time Frame: Baseline through 46 Months
Population: All participants who received at least one dose of ramucirumab and had evaluable immunogenicity samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - 750 mg Emibetuzumab | Part A - 2000 mg Emibetuzumab | Part B - Gastric | Part B - HCC | Part B - RCC | Part B - NSCLC
Number analyzed (Participants) | 3 | 3 | 16 | 44 | 15 | 15
Participants | 1 | 0 | 0 | 4 | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to 46 months
Description: All participants who received at least one dose of study drug. Gender specific events occurring only in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | Part A - 750 mg Emibetuzumab | Part A - 2000 mg Emibetuzumab | Part B - Gastric | Part B - HCC | Part B - RCC | Part B - NSCLC
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 3/16 | 4/45 | 1/15 | 1/15
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 4/16 | 19/45 | 5/15 | 3/15
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 15/16 | 45/45 | 15/15 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A - 750 mg Emibetuzumab (N=3) | Part A - 2000 mg Emibetuzumab (N=3) | Part B - Gastric (N=16) | Part B - HCC (N=45) | Part B - RCC (N=15) | Part B - NSCLC (N=15)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part A - 750 mg Emibetuzumab (N=3) | Part A - 2000 mg Emibetuzumab (N=3) | Part B - Gastric (N=16) | Part B - HCC (N=45) | Part B - RCC (N=15) | Part B - NSCLC (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 5 (5) | 7 (9) | 1 (1) | 2 (6)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 0 (0) | 7 (9) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (3)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 2 (2) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 9 (11) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (6) | 12 (14) | 3 (3) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 11 (12) | 2 (2) | 4 (6)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Gingival swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 8 (15) | 12 (16) | 4 (5) | 4 (6)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (4)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 6 (11) | 7 (8) | 1 (1) | 5 (7)
Asthenia (General disorders) | 1 (1) | 1 (1) | 5 (5) | 3 (4) | 1 (1) | 2 (2)
Breakthrough pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (3) | 11 (20) | 25 (34) | 6 (7) | 9 (13)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (4) | 1 (1) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 0 (0) | 6 (15) | 26 (38) | 5 (9) | 5 (9)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0)
Rubber sensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infected cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 2 (2)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 5 (5) | 2 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 6 (7) | 1 (2) | 1 (1)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 2 (4) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 2 (5) | 5 (5) | 1 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 3 (7) | 1 (1) | 0 (0)
Blood calcium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 1 (3)
Paracentesis (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (8) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 8 (8) | 11 (13) | 3 (4) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 6 (11) | 0 (0) | 2 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (5) | 13 (21) | 0 (0) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (11) | 0 (0) | 2 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (5) | 9 (15) | 2 (2) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 3 (3) | 3 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 5 (5) | 2 (2) | 3 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (4) | 2 (2) | 1 (1) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (4) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 4 (5) | 4 (4)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0/12 (0) | 0/34 (0) | 0/12 (0) | 1/9 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0/4 (0) | 0/11 (0) | 1/3 (1) | 0/6 (0)
Penile oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1/12 (1) | 0/34 (0) | 0/12 (0) | 0/9 (0)
Scrotal oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1/12 (1) | 0/34 (0) | 1/12 (1) | 0/9 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 3 (6) | 11 (12) | 4 (4) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 2 (5) | 12 (21) | 8 (9) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 7 (7) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 5 (5) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 11 (30) | 2 (2) | 2 (3)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release & can embargo communications regarding trial results for a period that is less than or equal to 30 days from the time submitted to sponsor for review. Sponsor can extend disclosure restriction for additional 60 days to protect intellectual property interests. If PI is unwilling to delay then PI shall remove the information that sponsor believes would jeopardize its IP interests

DOCUMENTS (2):
  • Study Protocol (2015-03-13): https://cdn.clinicaltrials.gov/large-docs/10/NCT02082210/Prot_000.pdf
  • Statistical Analysis Plan (2014-11-21): https://cdn.clinicaltrials.gov/large-docs/10/NCT02082210/SAP_001.pdf